CLINICAL TRIAL: NCT04031495
Title: Image Guidance for Improved Vessel Cannulation in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clear Guide Medical (Industry)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1R44HD096974-01 (NIH)
Record Dates: First submitted 2019-04-17; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Central Vein Cannulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: central vein cannulation — central vein cannulation

SUMMARY:
Feasibility Study This will be performed by an expert operator in Interventional Radiology who routinely performs CVC catheter placement, using appropriate pediatric human anatomy and vessel size, as well as real patient care scenarios.

DETAILED DESCRIPTION:
Phase I Feasibility Study This will be performed by an expert operator in Interventional Radiology who routinely performs CVC catheter placement, using appropriate pediatric human anatomy and vessel size, as well as real patient care scenarios. n=5 patients will be enrolled, and success would be 4 children (80%) successfully cannulated with a single pass using the P-SCENERGY.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients of weight between 5 and 25 kg requiring a central vein cannulation

Exclusion Criteria:

* none

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Successful Central Vein Cannulation | 1 day
  device enabled successful cannulation on the first pass showing feasibility to aid in cvcs

CONTACTS AND LOCATIONS:
Overall Officials: Karun Sharma, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No